CLINICAL TRIAL: NCT07327112
Title: Evaluation of the Anterior Tibialis Tendon Using Elastography in Patients With Hallux Valgus
Acronym: hallux valgus
Status: Not yet recruiting | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Recep Taşkin, Assistant Professor, Kastamonu University
Other Study IDs: KastamonuU123
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hallux Valgus Deformity; Elastography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hallux Valgus
- Control

SUMMARY:
To elucidate the relationship between changes in the mechanical properties of the tibialis anterior tendon and deformity in patients with hallux valgus, a case-control study is planned to quantitatively measure tendon stiffness using shear-wave elastography (SWE). Two groups will be compared: adults with radiographically confirmed hallux valgus (HVA (Hallux valgus angle) ≥15°) and age- and gender-matched healthy controls. The primary outcome is the elasticity modulus of the tibialis anterior tendon measured by SWE (kPa). Measurements will be performed using a high-frequency linear probe, with the probe positioned parallel to the tendon fibers and the foot in the standard ankle position, with three repetitions performed on each subject; the mean of stable frames will be used in the analysis. Secondary variables will be the relationships between tendon thickness/cross-sectional area, clinical angle parameters (HVA, IMA (intermetatarsal angle)), and functional scores. In the reliability sub-study, intra- and inter-observer ICC (Intraclass Correlation Coefficient), SEM (Standard Error of Measurement), and MDC (Minimal Detectable Change) will be calculated.

The sample size was calculated for a two-sample, two-tailed t-test with α=0.05 and 80% power assumptions, targeting a clinically meaningful medium-to-high effect size (Cohen d=0.60); at least 45 patients (45 with hallux valgus + 45 healthy) were planned. Parametric/non-parametric tests appropriate for the distribution and ANCOVA for potential confounders (age, gender, BMI, foot dominance) will be used in the analyses. The study is expected to objectively demonstrate whether tibialis anterior tendon stiffness changes in hallux valgus, thereby clarifying the muscle-tendon contributions to pathomechanics and laying the groundwork for targeted strategies in both conservative and surgical treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to provide written informed consent
* Compliance with procedures and ability to maintain standard position during measurement
* HV group: Weight-bearing radiograph showing HVA ≥15° (with IMA increase) - Control: no deformity, HVA <15°
* Selection of a single index foot in the same individual (highest HVA/symptomatic in HV; dominant in control)
* Availability or ability to obtain current radiographic measurements within the last 3 months

Exclusion Criteria:

* Previous foot/ankle surgery on the same lower extremity or significant trauma/fracture within the last 12 months
* Rheumatological/metabolic diseases (RA, spondyloarthritis, gout), neuropathy/peripheral vascular disease
* Drug/procedure affecting tendons: systemic or local corticosteroids within the last 6 months; fluoroquinolone use within the last 3 months
* Other significant foot deformity (advanced pes planus/cavus, hallux rigidus/varus) or professional intensive training (exclude or subgroup at your discretion)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visited the orthopedics outpatient clinic at Kastamonu Education and Research Hospital during the study period and were requested to undergo tibialis anterior tendon elastography examination
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Tibialis anterior tendon elasticity value | 1 Day
Determining the distal location of the anterior tibial tendon using ultrasound | 1 days

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available persistantly on 1.6.2026.
Access Criteria: Upon reasonable request principal investigator will share the data.